CLINICAL TRIAL: NCT06345638
Title: Sex Hormones and Inflammatory Biomarkers in Patients With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 854343
Record Dates: First submitted 2024-03-12; First posted 2024-04-03 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Females with SCD
- Males with SCD

SUMMARY:
This study aims to characterize sex differences in the pathophysiology of vaso-occlusive crises (VOC) occurring among individuals with sickle cell disease (SCD).

* The study will compare CRP and other biomarkers between females with SCD in the follicular phase of the menstrual cycle and males with SCD.
* The study will explore potential sex differences in biomarker changes between females and males with SCD during and following resolution of VOC.
* The study will compare neutrophil and platelet adhesion to the endothelium and real time fibrin deposition in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18-45
* Diagnosis of sickle cell disease
* current hospitalization for vaso-occlusive pain episode or current outpatient infusion at the recruiting sites
* Able to read and understand English
* Willing to comply with study procedures

Exclusion Criteria:

* Currently pregnant, pregnant within the last month, or seeking to become pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individual with sickle cell disease receiving care for vaso-occlusive pain episodes.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
C-reactive protein level | 1 month
  Serum level of hs-CRP

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Penn Medicine University City, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania